CLINICAL TRIAL: NCT06613022
Title: Effects of Instrument Assisted Soft Tissue Mobilization on Healthy Tissue Regarding Range of Motion and Grip Strength
Acronym: (IASTM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Marschner (Other)
Collaborators: Minot State University (Other)
Responsible Party: Sponsor-Investigator, Beth Marschner, Assistant Professor, Minot State University
Organization: Minot State University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2421
Record Dates: First submitted 2024-09-18; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Instrument Assisted Soft Tissue Mobilization; Range of Motion; Grip Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IASTM First (Experimental): This arm of the study received IASTM treatment on the first day and the wait/control on the second day of the study.
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization first Control second
- Wait/control First (Experimental): This arm of the study waited (was the control) on the first day and received IASTM treatment on the second day of the study.
  Interventions: Other: Control first Instrument Assisted Soft Tissue Mobilization second

INTERVENTIONS:
Other: Instrument Assisted Soft Tissue Mobilization first Control second — Instrument assisted soft tissue mobilization was utilized first on day one and wait-control was completed on second day.
  Arms: IASTM First
Other: Control first Instrument Assisted Soft Tissue Mobilization second — This intervention involved waiting for 20 minutes between pre-test and post-test on day one and having Instrument Assisted Soft Tissue Mobilization on day two.
  Arms: Wait/control First

SUMMARY:
The goal of this clinical trial is to study the effects of instrument assisted soft tissue mobilization (IASTM) in healthy adult volunteers. The main questions it aims to answer are:

* Does IASTM treatment have an effect on range of motion (ROM) as measured in the elbow, wrist and thumb?
* Does IASTM treatment have an effect on grip strength? Researchers will compare pre-test and post-test IASTM treatment intervention data to the pre-test and post-test data of the no treatment control intervention to see if IASTM works to change ROM and/or grip strength.

Participants will:

* Complete a questionnaire on medical history and injury background
* Have elbow, wrist, and thumb range of motion (ROM) measurements taken on both upper extremities using a goniometer
* Undergo grip strength testing using a JAMAR hand dynamometer in three positions on both upper extremities
* Be randomly assigned to either IASTM first treatment group or the wait/control first group
* Receive IASTM treatment techniques including application of emollient to the skin to reduce friction on the surface followed by scanning the forearm wrist flexors and wrist extensors and the biceps and triceps using the HG8-Scanner tool and then the concave tool corresponding to the size of the structure being treated will be used (HG6-Large Multi-Curve, HG5-Medium Multi-Curve, HG4-Small Multi-Curve) in each direction for a total treatment time of 20 minutes for both upper extremities in all listed areas.
* Simply wait for 20 minutes (the duration of time treatment with IASTM would require) when assigned to the control group.
* Complete elbow, wrist and thumb range of motion and grip strength measurement testing at the end of the first session.
* Return within fourteen days after the first session in order to undergo the opposite experience (IASTM first means wait/control second and vice versa).
* Undergo the same baseline pre-test measurements for range of motion and grip strength as the first session.
* Experience the opposite treatment group for the same time period as the first session.
* Undergo the post-test range of motion and grip strength testing at the end of the second session for data comparison.

DETAILED DESCRIPTION:
No further information to note than what is described in the summary or elsewhere

ELIGIBILITY:
Inclusion Criteria:

* A volunteer from a small regional university student body, faculty or staff may participate.

Exclusion Criteria:

* Acute spinal cord injury with neurological deficits
* Neurological disorders
* Acute upper extremity injury such as sprain or strain
* Any type of upper extremity fracture within the past 12 months
* Cervical disc pathology with radicular symptoms
* Use of blood thinning or clotting medications
* Known connective tissue disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Range of Motion | From baseline to end of session at one hour
  Bilateral elbow flexion and extension, wrist flexion, extension, ulnar deviation and radial deviation as well as thumb flexion, abduction and extension range of motion measurements were taken in sitting using a goniometer.
Grip Strength | From baseline to end of session at one hour
  Grip strength was assessed bilaterally using a JAMAR hand dynamometer. Three positions were tested. First the participant flexed their shoulder to 90 degrees with the elbow kept straight. Then the participant kept their arm down and their side with the elbow bent to 90 degrees. Finally the participant kept their arm down and straightened the elbow. Three trials were used for each position.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Marschner, DPT, Principal Investigator — Minot State University
Locations (1):
- Minot State University, Minot, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No
The individual participant data is not the main focus of this study. The overall findings of the study with the larger number of participants to look at the trend is what will be shared (presented or published). The IRB proposal for this study included confidentiality of each individual participant as that will be maintained, but the global findings are what will be shared after data analysis for comparison.